CLINICAL TRIAL: NCT00701662
Title: A Multicentre Study of Subcutaneous Immunoglobulin (SCIG) in Patients With Multifocal Motor Neuropathy (MMN)
Brief Title: A Study of Purified Human Antibodies Administered Subcutaneously to Patients With Multifocal Motor Neuropathy (MMN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1464; ZLB06_006CR (Other: CSL Behring); 2007-000710-37 (EudraCT Number)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-06

CONDITIONS: Multifocal Motor Neuropathy (MMN)
MeSH Terms: interventions — Vivaglobin; gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vivaglobin (Experimental): Vivaglobin® is a 16% (160 mg/mL) liquid formulation of human normal immunoglobulin for subcutaneous infusion. Subjects will receive weekly infusions of Vivaglobin® at a weekly dosage calculated based on previous intravenous immunoglobulin treatment (between 0.1 to 0.5 g/kg body weight per week).
  Interventions: Biological: Vivaglobin

INTERVENTIONS:
Biological: Vivaglobin
  Other Names: Human Normal Immunoglobulin

SUMMARY:
The objective of this study is to assess efficacy, safety, and convenience of purified human antibodies administered under the skin in the treatment of MMN patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented clinical diagnosis and electrophysiological evidence of MMN
* Patients who have previously responded to intravenous immunoglobulin (IVIG) and have been on stable treatment with IVIG for at least 12 weeks prior to screening
* Patients treated with the equivalent of ≥0.4g/kg body weight (bw) IVIG per month
* Provision of informed consent by patient

Exclusion Criteria:

* Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) concentration >2.5 times the upper normal limit (UNL)
* Creatinine concentration >1.5 times the UNL
* Known allergic reactions to blood products
* Any skin disease interfering with the assessment of injection site reactions
* Any other medical condition, which in the opinion of the investigator, might interfere with successful completion of the protocol
* Any condition likely to interfere with the evaluation of the study drug or satisfactory conduct of the trial
* Participation in a study with an investigational drug within three months prior to enrolment
* Patients treated with the equivalent of >2.0g/kg bw IVIG per month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Sturzenegger, MD, Principal Investigator — Inselspital, University Hospital of Bern; Bernd Kieseier, MD, Principal Investigator — Neurologische Klinik, Heinrich-Heine-University, Düsseldorf; Giancarlo Comi, MD, Principal Investigator — San Raffaele Hospital; Siraj Misbah, MD, Principal Investigator — Dept. Clinical Immunology, Oxford Radcliffe Hospitals
Locations (3):
- San Raffaele Hospital, Milan, Italy
- Inselspital, Bern, Switzerland
- Dept. Clinical Immunology, Oxford Radcliffe Hospitals, Oxford, United Kingdom

REFERENCES:
- [Result] Misbah S, et al. Efficacy and safety of subcutaneous immunoglobulin, Vivaglobin, in patients with multifocal motor neuropathy. Journal of Neurology 257(Suppl 1):S105-S106, 2010.
- [Result] Misbah SA, Baumann A, Fazio R, Dacci P, Schmidt DS, Burton J, Sturzenegger M. A smooth transition protocol for patients with multifocal motor neuropathy going from intravenous to subcutaneous immunoglobulin therapy: an open-label proof-of-concept study. J Peripher Nerv Syst. 2011 Jun;16(2):92-7. doi: 10.1111/j.1529-8027.2011.00330.x. PMID 21692906

RESULTS

PARTICIPANT FLOW:
Groups:
- Vivaglobin: Human normal immunoglobulin, 0.1 to 0.5 g/kg body weight per week.
Period: Overall Study
Arm/Group | Vivaglobin
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.78)
Age, Customized [Number; unit: participants]
  > 18 to < 65 years | 5
  >= 65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Muscle Strength
Description: The change in Medical Research Council (MRC) score was determined at week 24 compared to baseline using descriptive statistics and nonparametric, two-sided 95% confidence intervals based on the Hodges-Lehmann method. Data for one of the eight subjects was from week 13 as week 24 data were not available.
  The 200-point MRC sum score is the sum of scores for 20 bilateral (left and right side) muscle groups, each rated between 0 (no movement) to 5 (normal movement/power). A higher MRC sum score indicates greater muscle contraction/limb movement. Positive values for change in MRC sum score indicate improvement, with a more positive value indicating greater muscle contraction/ limb movement compared with the value at baseline.
Time Frame: Baseline to week 24
Population: The Intention-to-Treat (ITT) data set comprised all patients treated with the study drug who had at least one post-baseline measurement for muscle strength.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale | 0.4 (5.07) [-4.50 to 5.00]

2. Secondary Outcome: Change From Baseline to Week 24 in Disability
Description: The change in disability score was determined at week 24 compared to baseline using descriptive statistics and nonparametric two-sided 95% confidence intervals based on the Hodges-Lehmann method. Data for one of the eight subjects was from week 13 as week 24 data were not available.
  Disability was measured using a modified Guy's Neurological Disability Scale, which comprises subscales for upper and lower limb disability. Both subscales comprise 6 grades, numbered from 0 (no upper limb problem/walking is not affected) to 5 (unable to use either arm for any purposeful movements/usually uses a wheelchair indoors). The disability score is calculated as the sum of both subscales, resulting in a score ranging from 0 to 10. A higher disability score indicates greater disability. Negative values for change in disability score indicate improvement, with a more negative value indicating greater improvement compared with the value at baseline.
Time Frame: Baseline to week 24
Population: The analysis population comprised the subjects in the ITT data set (ie, all patients treated with the study drug) who had at least one post-baseline value (and if necessary a baseline value).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale | 0.1 (1.13) [-1.00 to 1.00]

3. Secondary Outcome: Mean Disability Score at Baseline and Week 24
Description: Disability was measured using a modified Guy's Neurological Disability Scale, which comprises subscales for upper and lower limb disability. Both subscales comprise 6 grades, numbered from 0 (no upper limb problem/walking is not affected) to 5 (unable to use either arm for any purposeful movements/usually uses a wheelchair indoors). The disability score is calculated as the sum of both subscales, resulting in a score ranging from 0 to 10. A higher disability score indicates greater disability.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale
  Disability score at baseline (n = 8) | 2.0 [1 to 3]
  Disability score at week 24 (n = 7) | 1.9 [1 to 3]

4. Secondary Outcome: Change From Baseline to the Completion Visit in Motor Function
Description: The change in motor function was determined at the completion visit compared to baseline using descriptive statistics and nonparametric two-sided 95% confidence intervals based on the Hodges-Lehmann method.
  For each patient, four specific tasks were defined according to his/her weakened muscle group. The patient had to grade each of the tasks on a 5-point scale ranging from 0 (normal function) to 4 (not possible). The overall motor function score was calculated as the sum of the 4 grades, resulting in a score ranging from 0 (optimal) to 16 (worst). The baseline motor function score was calculated as the mean of the patient's assessments at Screening and Week 1. Negative values for change in motor function score indicate improvement, with a more negative value indicating greater improvement compared with the value at baseline.
Time Frame: Baseline to the completion visit (up to week 25)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale | 0.4 (1.94) [-1.50 to 0.75]

5. Primary Outcome: Mean Overall MRC Score at Baseline and Week 24
Description: The 200-point MRC sum score is the sum of scores for 20 bilateral (left and right side) muscle groups, each rated between 0 (no movement) to 5 (normal movement/power). A higher MRC sum score indicates greater muscle contraction/limb movement.
Time Frame: Baseline and week 24
Population: The ITT data set comprised all patients treated with the study drug who had at least one post-baseline measurement for muscle strength.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale
  MRC score at baseline (n = 8) | 178.3 [149 to 197]
  MRC score at week 24 (n = 7) | 184.3 [171 to 198]

6. Secondary Outcome: Mean Motor Function Score at Screening and Week 25
Description: For each patient, four specific tasks were defined according to his/her weakened muscle group. The patient had to grade each of the tasks on a 5-point scale ranging from 0 (normal function) to 4 (not possible). The overall motor function score was calculated as the sum of the 4 grades, resulting in a score ranging from 0 (optimal) to 16 (worst).
Time Frame: Screening and week 25
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
score on a scale
  Motor function score at screening (n = 8) | 5.5 [0 to 8]
  Motor function score at week 25 (n = 7) | 4.6 [0 to 8]

7. Secondary Outcome: Health-Related Quality of Life at Baseline and Week 25
Description: Assessed using a questionnaire on patients' satisfaction with current immunoglobulin G (IgG) treatment, treatment at home, and treatment at the hospital/doctor's office. The questions were answered by choosing a number between 1 (extremely good) and 7 (extremely bad).
  Note: No patients received IgG treatment at the hospital/doctor's office at Week 25.
Time Frame: At baseline and week 25
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
units on a scale
  Current treatment, baseline (n = 8) | 2.6 (1.06) [1 to 4]
  Current treatment, week 25 (n = 7) | 1.3 (0.49) [1 to 2]
  At home, baseline (n = 3) | 1.0 (0.00) [1 to 1]
  At home, week 25 (n = 7) | 1.1 (0.38) [1 to 2]
  In the hospital/doctor's office, baseline (n = 7) | 2.9 (1.57) [1 to 5]

8. Secondary Outcome: Treatment Satisfaction at Baseline and Week 25
Description: Treatment satisfaction was assessed using the Life Quality Index, which comprises 15 items rated on a 7-point scale (1 = worst rating, 7 = best rating) with a possible maximum score of 105. The highest score indicates the highest satisfaction with the impact of treatment on social factors. The 15 items were summarized to 4 scales: treatment interference, therapy-related problems, therapy setting, and treatment costs. The raw scores for these scales were transformed to a score ranging from 0 to 100, with 100 being the best score achievable.
Time Frame: At baseline and week 25
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
units on a scale
  Treatment interference, baseline (n = 8) | 60.76 (25.827) [8.3 to 97.2]
  Treatment interference, week 25 (n = 6) | 91.67 (9.780) [75.0 to 100.0]
  Therapy-related problems, baseline (n = 8) | 70.30 (27.055) [8.3 to 91.7]
  Therapy-related problems, week 25 (n = 7) | 89.29 (14.402) [66.7 to 100.0]
  Therapy setting, baseline (n = 8) | 75.01 (33.844) [5.6 to 100.0]
  Therapy setting, week 25 (n = 6) | 96.28 (6.743) [83.3 to 100.0]
  Treatment costs, baseline (n = 8) | 70.84 (34.498) [0.0 to 100.0]
  Treatment costs, week 25 (n = 6) | 86.10 (19.486) [50.0 to 100.0]

9. Secondary Outcome: Overall Health Status at Baseline and Week 25
Description: Overall Health Status was assessed using a Visual Analogue Scale (VAS). Patients were asked to rate their overall health status by placing a mark on a 100 mm VAS, with 0 being the worst imaginable state and 100 being the best imaginable state.
Time Frame: Baseline and week 25
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
units on a scale
  Baseline (n = 8) | 72.1 (15.38) [52 to 96]
  Week 25 (n = 7) | 73.9 (14.67) [50 to 98]

10. Secondary Outcome: Number of Patients With Adverse Events (AEs) by Severity and Relatedness
Description: Included all AEs that occurred during the entire study period.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to Week 25
Population: The safety data set (SDS) comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
participants
  All AEs | 4
  Mild AEs | 3
  Moderate AEs | 2
  Severe AEs | 0
  Not related AEs | 4
  Possibly related AEs | 0
  Probably related AEs | 0
  Related AEs | 1

11. Secondary Outcome: Rate of AEs by Severity and Relatedness
Description: The rate was the number of AEs over the number of infusions administered. Included all AEs that occurred during the entire study period.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to Week 25
Population: The SDS comprised all treated patients.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
Number analyzed (Infusions) | 183
AEs per infusion
  All AEs | 0.104
  Mild AEs | 0.093
  Moderate AEs | 0.011
  Severe AEs | 0.000
  Not related AEs | 0.038
  Possibly related AEs | 0.000
  Probably related AEs | 0.000
  Related AEs | 0.066

12. Secondary Outcome: Number of Patients With Local/Injection Site Reactions
Description: All AEs arising from local/injection site reactions.
Time Frame: For the duration of the study, up to Week 25
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
participants
  Total | 1
  Injection site oedema | 1
  Injection site pruritis | 1
  Skin reaction | 1

13. Secondary Outcome: Number of Patients With Clinically Relevant Changes in Laboratory Parameters
Description: Laboratory parameters included hematology, serum chemistry, and urinalysis parameters.
Time Frame: Baseline to Week 25
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
participants | 0

14. Secondary Outcome: Number of Patients With Clinically Relevant Changes in Vital Signs
Description: Vital signs included heart rate, systolic blood pressure, diastolic blood pressure, and body temperature.
Time Frame: Baseline to Week 25
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
participants | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to Week 25.
Description: The SDS comprised all treated patients. "General disorders" were collected under the Medical Dictionary for Regulatory Activities System organ class (MedDRA SOC) General disorders and administration site conditions.
Arm/Group | Vivaglobin
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaglobin (N=8)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Injection-site oedema (General disorders) | 1 (4)
Injection-site pruritus (General disorders) | 1 (4)
Influenza (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Hemicephalalgia (Nervous system disorders) | 1 (1)
Multifocal motor neuropathy (Nervous system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.